CLINICAL TRIAL: NCT00767689
Title: A Randomized Trial to Determine if Vitamin B6 Can Prevent Hand and Foot Syndrome in Cancer Patients Treated With Capecitabine Chemotherapy
Brief Title: Vitamin B6 Can Prevent Hand and Foot Syndrome in Cancer Patients Capecitabine Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: incomplete enrollment
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Pamela Gonzalez Sr Director Clinical Research Office, Dir Clinical Research Office, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-069
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hand and Foot Syndrome
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Vitamin B 6; Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin B6 (Experimental): patient receiving xeloda and vitamin B6
  Interventions: Drug: Vitamin B 6
- 2 placebo (Placebo Comparator): patient receiving xeloda and placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin B 6 — vitamin b6 100 mg po daily
  Other Names: pyridoxine
  Arms: vitamin B6
Drug: placebo — placebo is given in the placebo arm
  Arms: 2 placebo

SUMMARY:
Capecitabine (Xeloda) a drug in cancer therapy. Its use is limited often by its toxicities. This study is asking if vitamin B6 can prevent one of the common toxicities of xeloda which is numbness and/or rash of the hands and feet, a condition called Hand and Foot syndrome. patients , starting capecitabine chemotherapy for their cancer, will participate in this study at John H. Stroger Jr. Hospital of Cook County. They will be randomized to receive either vitamin B6 or a placebo. investigators and patients will be blinded to the intervention.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled trial, with randomly assignment of eligible patients who were treated with capecitabine to receive either daily pyridoxine 100 mg or placebo along with their capecitabine-containing chemotherapy regimen. Patients were observed during the first 4 cycles of capecitabine treatment. The primary endpoint was the incidence and grade of Hand-Foot Syndrome (HFS) that occurred in both study arms.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient starting capecitabine-containing chemotherapy
* Has never had capecitabine before
* Performance status 0-2 using the ECOG classification
* Life expectancy more than 6 months
* Agreed to stop any vitamin supplements, apart from vitamin D.
* Liver function studies including AST/ALT within 3x upper limit of normal
* Signed informed consent must be obtained from participating individuals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-03-21 (Actual); Primary Completion 2009-03-18 (Actual); Study Completion 2010-03-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Hand-Foot Syndrome (HFS) | 1 year
  Incidence of HFS based on CTCTAE adverse event table

SECONDARY OUTCOMES:
Grade of Hand-Foot Syndrome (HFS) | 1 year
  Grading of HFS: Grade 1, Grade 2, Grade 3 per NCI CTCTAE V 3

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lad, MD, Study Director — Cook County Health Oncology NCORP; Susan McDunn, MD, Principal Investigator — Cook County Health
Locations (1):
- John H stroger Jr hospital of cook county, Chicago, Illinois, United States